CLINICAL TRIAL: NCT05167370
Title: High Dose Chemotherapy With Amifostine and Autologous Stem Cell Transplantation for High Risk Relapsed Pediatric Solid Tumors and Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as recommended by the DSMB due to inability to meet enrollment goals within the time frame allotted (target of 25 patients over 5 years).
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amifostine
Record Dates: First submitted 2012-08-01; First posted 2021-12-22 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumors; Brain Tumors
Keywords: Solid Tumors; Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amifostine (Experimental)
  Interventions: Drug: Amifostine

INTERVENTIONS:
Drug: Amifostine — Amifostine (Ethyol) 1125 mg/m2 will be given intravenously daily over 5 minutes starting 30 minutes prior to chemotherapy (melphalan or thiotepa) on days -5, -4, -3, -2, and on day -1 twenty four hours after prior dose of amifostine.
  Other Names: Ethyol

SUMMARY:
This is a study of amifostine to determine how effective it is in the reduction of infection in a high dose chemotherapy regimen with autologous stem cell rescue in children with high risk, relapsed or refractory pediatric solid tumors.

DETAILED DESCRIPTION:
Autologous stem cell transplant (ASCT) permits chemotherapy dose-escalation to exploit the steep dose-response of solid tumors to alkylating agents. Although ASCT regimens have activity in some high risk pediatric solid tumors, non-hematological regimen-related morbidity and mortality are major barriers to additional dose escalation. We hypothesized that the chemoprotectant amifostine (Ethyol®) would reduce the toxicity of ASCT without compromising anti-tumor efficacy. This is a study of amifostine at 1125 mg/m2 to determine the efficacy of it's chemoprotection in the reduction of bacteremia in a high dose busulfan, melphalan and thiotepa chemotherapy regimen with autologous stem cell rescue in children with high risk, relapsed or refractory pediatric solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* High risk Ewing's Sarcoma Family Tumors (ESFT) including Ewing's Sarcoma, Askin's tumor, peripheral PNET
* High risk desmoplastic small round cell tumors (DSRCT)
* Relapsed Wilm's tumor, diffuse anaplastic Wilm's tumor
* High risk brain tumors including PNET/Medulloblastomas/germinomas
* Relapsed germ cell tumors
* Metastatic or relapsed rhabdoid tumors
* Other relapsed/refractory pediatric embryonal tumors
* Less than 30 years of age
* Performance >= 50%
* Cancer Diagnosis verification and staging
* Disease Response and Recovery
* Adequate Organ Function (Renal, Liver, Cardiac)

Exclusion Criteria:

* Uncontrolled Infection
* Pregnancy or Breastfeeding (For Females)
* Disease Progression
* Uncontrolled Intercurrent Illness
* HIV Positive
* Receiving other Investigational Agents
* Amifostine Allergy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2011-04-29 (Actual); Study Completion 2012-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonata Jodele, MD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amifostine
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amifostine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bacteriemia in a High Dose Busulfan, Melphalan and Thiotepa Chemotherapy Regimen With Autologous Peripheral Blood Stem Cell Rescue in Patients With High Risk and Relapsed or Refractory Pediatric Solid Tumors
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amifostine
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Through 30 days after the end of protocol therapy
Arm/Group | Amifostine
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amifostine (N=2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Disease Progression (General disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No